CLINICAL TRIAL: NCT03727958
Title: Simultaneous Coronary Artery Evaluation and Lung Cancer Screening With a New Ultrafast-low-dose Computed Tomography Protocol: A Pilot Randomized Trial
Brief Title: Simultaneous Coronary Artery Evaluation and Lung Cancer CT Screening
Acronym: SIMULTANEOUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/D/789
Record Dates: First submitted 2018-10-28; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: HEAVY SMOKING

STUDY DESIGN:
Intervention Model Description: Current or former heavy smoker subjects with suspected or known coronary artery disease will be randomized to undergo CT assessment of both coronary arteries and thoracic area for simultaneous coronary artery and lung cancer screening
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung and coronary CT assessment (Active Comparator): Subjects will undergo simultaneous CT assessment of both coronary arteries and thoracic area
  Interventions: Diagnostic Test: Lung and coronary CT assessment
- Coronary CT assessment (Active Comparator): Subjects will undergo CT assessment of coronary arteries only
  Interventions: Diagnostic Test: Coronary CT assessment

INTERVENTIONS:
Diagnostic Test: Lung and coronary CT assessment — Subjects will undergo simultaneous coronary arteries and thoracic CT assessment
  Arms: Lung and coronary CT assessment
Diagnostic Test: Coronary CT assessment — Subjects will undergo coronary arteries CT assessment only
  Arms: Coronary CT assessment

SUMMARY:
Cardiac computed tomography (CT) is often performed in patients who are at high risk for lung cancer in whom screening is currently recommended. This pilot randomized study will test the feasibility, safety and diagnostic ability of a novel ultra-low-dose CT protocol that allows concomitant coronary artery evaluation and lung screening. Current or former heavy smoker subjects with suspected or known coronary artery disease will be randomized to undergo CT assessment of either thoracic area only or both coronary arteries and thoracic area. Primary end-points will be the effective contrast and radiation doses.

DETAILED DESCRIPTION:
Cardiac computed tomography (CT) scan is an ideal diagnostic tool for identifying coronary artery disease in patients with low or intermediate risk. In recent years, cardiac CT is being often performed in patients who are at high risk either for coronary artery disease or lung cancer. The update edition of the National Institute for Health and Care Excellence (NICE) guidelines recommends cardiac CT as the first-line diagnostic tool for patients with new-onset chest pain due to suspected coronary artery disease. Also, symptomatic patients with known coronary artery disease and previous percutaneous coronary intervention who have an unclear stress test but whose presentation suggests a high likelihood of having an in-stent restenosis or a 'de novo' stenosis might benefit from cardiac CT. In 2014, the U.S. Preventive Services Task Force recommended annual lung cancer screening with ultra-low dose computed tomography for current and former heavy smokers aged 55 to 80 years. Indeed, lung cancer screening in patients with suspected or known coronary artery disease undergoing cardiac CT may provide the opportunity to implement recommendation for lung cancer screening in clinical practice.This pilot randomized study will test the feasibility, safety and diagnostic ability of a novel ultra-low-dose CT protocol that allows concomitant coronary artery evaluation and lung screening. Current or former heavy smoker subjects with suspected or known coronary artery disease will be randomized to undergo CT assessment of either thoracic area only or both coronary arteries and thoracic area. Primary end-points will be the effective contrast and radiation doses.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic subjects with effort-induced or typical chest pain
* High probability of coronary artery disease
* Known coronary artery disease
* Willing to participate to the study
* Informed consent to undergo CT scan

Exclusion Criteria:

* Contraindications to iodinated contrast such as allergies and chronic kidney failure
* Any suspicion of pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of computed tomography as measured by effective radiation dose (as measured in mSv) | Through study completion, an average of 2 months
  Measurement of the effective radiation dose (as measured in mSv) at time of computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaudio C, Tanzilli A, Mei M, Moretti A, Barilla F, Varveri A, Paravati V, Tanzilli G, Ciccaglioni A, Strano S, Pellegrini M, Barillari P, Pelliccia F. Concomitant screening of coronary artery disease and lung cancer with a new ultrafast-low-dose Computed Tomography protocol: A pilot randomised trial. Sci Rep. 2019 Sep 25;9(1):13872. doi: 10.1038/s41598-019-50407-6. PMID 31554878